CLINICAL TRIAL: NCT01018680
Title: A Randomized, Placebo-Controlled Trial of Duloxetine Added to Nonsteroidal Anti-inflammatory Drugs in Patients With Knee Pain Due to Osteoarthritis Who Have Had Suboptimal Response to Nonsteroidal Anti-inflammatory Drug Treatment.
Brief Title: A Study Comparing Duloxetine Versus Placebo in Patients Taking a Nonsteroidal Anti-inflammatory Drug (NSAID) for Knee Pain Due to Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12909; F1J-US-HMGL (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis Knee Pain
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — 30 milligrams (mg) taken by mouth, once daily for 1 week, followed by 60 to 120 mg taken by mouth, once daily for 9 weeks.
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine
Drug: Placebo — Taken by mouth, once daily for 10 weeks
  Arms: Placebo

SUMMARY:
The study will test the hypothesis that, in patients with knee pain due to osteoarthritis (OA) who are taking nonsteroidal anti-inflammatory drugs (NSAIDs) but still have significant knee pain, duloxetine 60 to 120 milligrams (mg) daily for 10 weeks will provide additional reduction in pain.

DETAILED DESCRIPTION:
Duloxetine has been studied in pain due to osteoarthritis (OA) in 2 previous placebo controlled clinical trials. In clinical practice, when nonsteroidal anti-inflammatory drugs (NSAIDs) are ineffective in reducing pain due to OA, clinicians often add a second agent without discontinuing NSAIDs. In this study, we will investigate whether adding duloxetine to NSAIDs provides additional pain relief and functional improvement in patients with knee pain due to OA.

ELIGIBILITY:
Inclusion Criteria:

* Present with knee pain due to osteoarthritis (OA) based on OA clinical and radiographic diagnostic criteria.
* Knee Pain for > 14 days of each month for the 3 months directly preceding study entry.
* Taking nonsteroidal anti-inflammatory drugs (NSAIDs) for knee pain due to OA on most days in the 3 months immediately preceding study entry.

Exclusion Criteria:

* History of intolerance or nonresponsiveness to an adequate trial of duloxetine used for any indication, in the opinion of the investigator.
* Previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder.
* Have major depressive disorder (MDD) as determined using depression module of the Mini International Neuropsychiatric Interview (MINI).
* Judged clinically by the investigator to be at suicidal risk by examination or using the Columbia Suicide Severity Rating Scale (C-SSRS).
* History of substance abuse or dependence within the past year, excluding nicotine and caffeine.
* Positive urine drug screen for any substance of abuse or excluded medication.
* Opioid dependent in the opinion of the investigator, taking opioids more than 3 days a week, or unwilling to discontinue opioids during the study period.
* Known hypersensitivity to duloxetine or its inactive ingredients.
* History of intolerance or hypersensitivity to NSAIDS, Cyclooxygenase (COX-2) inhibitors, or proton pump inhibitors.
* History of peptic ulcer disease, bleeding disorder, gastrointestinal bleeding, or any abnormal bleeding.
* Baseline hemoglobin measurement of <11 grams per deciliter (g/dL) for males, or <10 g/dL for females.
* Serious or unstable cardiovascular, hepatic, renal, metabolic, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or any other medical or psychiatric condition that would compromise participation or be likely to lead to hospitalization or a change in medication during the course of the study.
* Uncorrected thyroid disease, uncontrolled narrow-angle glaucoma, uncontrolled or poorly controlled hypertension, or history of seizures.
* Active liver injury (such as hepatitis) or any degree of hepatic insufficiency (Child-Pugh Class C).
* Frequent falls that could result in hospitalization or could compromise response to treatment.
* Confounding painful condition that may interfere with assessment of the index knee.
* Chronic widespread pain affecting all four quadrants of the body, or diagnosis of fibromyalgia.
* Received intra-articular hyaluronate (Synvisc), steroids, joint lavage, or other invasive therapies to the knee in the past 6 months.
* Arthroscopy of the index knee within the past year or joint replacement of the index knee at anytime.
* Diagnosis of inflammatory arthritis (that is, rheumatoid arthritis, psoriatic arthritis, reactive arthritis, ankylosing spondylitis, etc.) or an autoimmune disorder (excluding inactive Hashimoto's thyroiditis).
* Prior synovial fluid analysis showing a white blood cell count greater than or equal to 2000 cubic millimeters (mm^3) that is indicative of a diagnosis other than OA, or have a history of gout or pseudogout.
* Radiographic evidence of end-stage (bone on bone) OA in either knee.
* Knee replacement surgery planned within the next 6 months.
* Nonambulatory or requiring the use of crutches, a walker, or more than 1 cane.
* Body mass index (BMI) >40.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- United States (32):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildomar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boulder, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cromwell, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Sterling, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pasadena, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wheaton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fall River, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Weymouth, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manlius, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duncansville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warwick, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Germán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

REFERENCES:
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Westfall PH, Krishen A. Optimally weighted, fixed sequence and gatekeeper multiple testing procedures. J Stat Plann Infer. 2001;99(1):25-40.
- [Derived] Yue L, Wang J, Enomoto H, Fujikoshi S, Alev L, Cheng YY, Skljarevski V. The Clinical Relevance of Pain Severity Changes: Is There Any Difference Between Asian and Caucasian Patients With Osteoarthritis Pain? Pain Pract. 2020 Feb;20(2):129-137. doi: 10.1111/papr.12835. Epub 2019 Nov 20. PMID 31505082
- [Derived] Risser RC, Hochberg MC, Gaynor PJ, D'Souza DN, Frakes EP. Responsiveness of the Intermittent and Constant Osteoarthritis Pain (ICOAP) scale in a trial of duloxetine for treatment of osteoarthritis knee pain. Osteoarthritis Cartilage. 2013 May;21(5):691-4. doi: 10.1016/j.joca.2013.02.007. Epub 2013 Feb 26. PMID 23485934
- [Derived] Frakes EP, Risser RC, Ball TD, Hochberg MC, Wohlreich MM. Duloxetine added to oral nonsteroidal anti-inflammatory drugs for treatment of knee pain due to osteoarthritis: results of a randomized, double-blind, placebo-controlled trial. Curr Med Res Opin. 2011 Dec;27(12):2361-72. doi: 10.1185/03007995.2011.633502. Epub 2011 Nov 9. PMID 22017192

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo by mouth, once daily for 10 weeks.
- Duloxetine: Participants initially received 30 milligrams (mg) duloxetine by mouth, once daily for 1 week, followed by 60 mg by mouth, once daily thereafter. At end of 3 weeks, participants with a weekly mean 24-hour average pain value ≥4 in week preceding their visit had their dose escalated up to 120 mg by mouth, once daily until Week 10.
Period: Overall Study
Arm/Group | Placebo | Duloxetine
Started | 260 | 264
Completed | 199 | 189
Not Completed | 61 | 75
Not completed — Adverse Event | 23 | 40
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Protocol Violation | 5 | 8
Not completed — Sponsor Decision | 6 | 7
Not completed — Lack of Efficacy | 8 | 2
Not completed — Lost to Follow-up | 5 | 3
Not completed — Entry Criteria Not Met | 1 | 4
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Duloxetine | Total
Number analyzed (Participants) | 260 | 264 | 524
Age Continuous [Mean (Standard Deviation); unit: years] | 60.32 (9.17) | 61.63 (9.24) | 60.98 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 152 | 299
  Male | 113 | 112 | 225
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 38 | 84
  White | 206 | 218 | 424
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 260 | 264 | 524
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 90.78 (17.49) | 90.41 (18.13) | 90.59 (17.80)
Weekly 24-Hour Average Pain Rating [Mean (Standard Deviation); unit: units on a scale] — The weekly 24-hour average pain rating was calculated from the participant's daily 24-hour average pain ratings made on an 11-point numeric rating scale, with scores from 0 (indicating "no pain") to 10 (indicating "the worst possible pain") from the week ending at the day of randomization.
  units on a scale | 6.36 (1.41) | 6.27 (1.41) | 6.32 (1.41)
Brief Pain Inventory-Severity (BPI-S) Average Pain [Mean (Standard Deviation); unit: units on a scale] — The BPI-S is a self-reported scale measuring severity of pain. Severity score ranges from 0 (no pain) to 10 (severe pain) assessing average pain in past 24 hours.
  units on a scale | 6.24 (1.51) | 6.09 (1.58) | 6.16 (1.54)
Patient Global Assessment of Illness (PGAI) [Mean (Standard Deviation); unit: units on a scale] — The PGAI is a participant-rated measure of the severity of osteoarthritis (OA) of the knee the participant has experienced in the past week as indicated on an 11-point numeric rating scale, with scores ranging from 0 to 10, where greater numbers reflect greater severity.
  units on a scale | 6.95 (1.50) | 6.93 (1.49) | 6.94 (1.49)
Western Ontario and McMaster Universities Index of Osteoarthritis Physical Function Score [Mean (Standard Deviation); unit: units on a scale] — The Western Ontario and McMaster Universities Index of Osteoarthritis Physical Function Score (WOMAC; Bellamy et al. 1988) is a self-administered, participant-centered health status questionnaire used to capture the elements of pain, stiffness, and physical disability in participants with osteoarthritis (OA) of the knee and/or hip. The physical function index has 17 questions. Each question uses a 5-point numeric rating scale ranging from 0 (no difficulty) to 4 (extreme difficulty). Physical function scores range from 0 to 68, where higher scores indicate greater impairment.
  units on a scale | 37.51 (9.39) | 37.40 (10.10) | 37.45 (9.74)
Duration of Osteoarthritis (OA) Pain [Mean (Standard Deviation); unit: years] | 9.19 (8.92) | 9.79 (8.88) | 9.49 (8.90)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Mean of the 24-Hour Average Pain Score at 8 Weeks
Description: The weekly mean 24-hour average pain score was calculated from the participant's daily 24-hour average pain ratings using an 11-point numeric rating scale, with scores from 0 (indicating "no pain") to 10 (indicating "the worst possible pain"). The Least Squares Mean estimates were adjusted for baseline, treatment, investigator (pooled), week, treatment*week, and baseline*week.
Time Frame: Baseline, 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline weekly mean 24-hour average pain value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 255 | 259
units on a scale | -1.55 (0.11) | -2.46 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Using a 1:1 ratio of allocation to treatment, a 2-tailed 0.05 level of significance and 80% power, 253 participants per arm had been estimated to be adequate to assess an effect size of 0.25, based on a 2-sample Student's t-test. This derived estimate was increased slightly to 261 participants per arm to account for extremely early discontinuation that would have led to exclusion from the efficacy analysis in a small number of participants (approximately 3%); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.91

2. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at 8 Weeks
Description: A scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). The Least Squares Mean estimates were adjusted for baseline value of Patient Global Impression of Severity (PGI-S), treatment, investigator (pooled), visit, and treatment*visit. The PGI-S measures participant's perception of severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (extremely ill).
Time Frame: 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline PGI-S rating and at least 1 post-baseline PGI-I rating were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 254 | 254
units on a scale | 2.93 (0.09) | 2.33 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — First gated secondary outcome measure. Gatekeeper strategy (Westfall and Krishen 2001) controlled experiment-wise type I error for 2 secondary outcomes with sequential comparisons of treatments until outcome failed to be significant (p>0.05); In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.59

3. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC) Pain, Stiffness, and Physical Function Subscale Scores at 8 Weeks
Description: Self-administered questionnaire captures elements of pain, stiffness, and physical disability in participants with osteoarthritis of the knee and/or hip. Index has 24 questions (5 on pain, 2 on stiffness, 17 on physical function). Each question uses a 5-point numeric rating scale ranging from 0 (none) to 4 (extreme). Pain scores range: 0 to 20. Stiffness scores range: 0 to 8. Physical function scores range: 0 to 68. Higher scores=greater impairment. Least Squares Mean estimates were adjusted for baseline value, treatment, investigator (pooled), visit, treatment*visit, and baseline value*visit.
Time Frame: Baseline, 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline WOMAC value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 256 | 258
units on a scale
  WOMAC Physical Disability Score (n=253, 251) | -10.25 (0.82) | -15.09 (0.81)
  WOMAC Pain Score | -3.13 (0.24) | -4.41 (0.23)
  WOMAC Stiffness Score | -1.45 (0.12) | -1.88 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — WOMAC Physical Disability Score p-value. Second gated secondary outcome measure. Gatekeeper strategy controlled experiment-wise type I error for 2 secondary outcomes with sequential treatment comparisons until outcome failed significance (p>0.05); In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -4.84
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the WOMAC Pain Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -1.28
Statistical Analysis 3: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — This is the p-value for WOMAC Stiffness Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.42

4. Secondary Outcome: Change From Baseline in the Weekly Mean of the 24-Hour Night Pain and Worst Pain Scores at 8 Weeks
Description: Weekly mean 24-hour night pain and worst pain values are calculated from the participant's daily assessments of pain at night and worst pain during the previous 24 hours on an 11-point numeric rating scale, with scores from 0 (indicating "no pain") to 10 (indicating "the worst possible pain"). The Least Squares Mean estimates were adjusted for baseline value, treatment, investigator (pooled), week, treatment*week, and baseline*week.
Time Frame: Baseline, 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline night/worst pain value and at least 1 post-baseline weekly mean 24-hour night/worst pain value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 253 | 259
units on a scale
  Night Pain Intensity | -1.46 (0.11) | -2.26 (0.11)
  Worst Pain Intensity | -1.58 (0.13) | -2.61 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for Night Pain Intensity. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.80
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for Worst Pain Intensity. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -1.03

5. Secondary Outcome: Change From Baseline in the Brief Pain Inventory Severity and Interference Scores (BPI-S/BPI-I) Scores at 8 Weeks
Description: Measures pain severity and pain interference with function. Severity scores: 0 (no pain) to 10 (severe pain) on each question. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Mean interference is the average across the 7 interference items. The Least Squares Mean estimates were adjusted for baseline value, treatment, investigator (pooled), visit, treatment*visit, and baseline*visit.
Time Frame: Baseline, 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline BPI-S/BPI-I value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 256 | 258
units on a scale
  BPI-S for Worst Pain | -1.87 (0.17) | -2.94 (0.17)
  BPI-S for Least Pain | -1.44 (0.14) | -2.14 (0.14)
  BPI-S for Average Pain | -1.78 (0.15) | -2.73 (0.15)
  BPI-S for Pain Right Now | -2.03 (0.16) | -2.74 (0.16)
  BPI-I for General Activity | -1.79 (0.17) | -2.76 (0.16)
  BPI-I for Mood | -1.80 (0.15) | -2.52 (0.15)
  BPI-I for Walking Ability | -1.85 (0.17) | -2.80 (0.17)
  BPI-I for Normal Work | -1.92 (0.17) | -2.77 (0.17)
  BPI-I for Relations with Others (n=255, 258) | -1.25 (0.14) | -1.94 (0.14)
  BPI-I for Sleep | -2.01 (0.14) | -2.69 (0.14)
  BPI-I for Enjoyment of Life | -1.89 (0.17) | -2.66 (0.17)
  BPI-I for Mean Interference Score | -1.77 (0.14) | -2.60 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-S for Worst Pain. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -1.08
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-S for Least Pain. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.70
Statistical Analysis 3: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-S for Average Pain. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.95
Statistical Analysis 4: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-S for Pain Right Now. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.71
Statistical Analysis 5: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for General Activity. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.97
Statistical Analysis 6: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for Mood. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.72
Statistical Analysis 7: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for Walking Ability. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.95
Statistical Analysis 8: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for Normal Work. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.85
Statistical Analysis 9: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for Relations with Others. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.69
Statistical Analysis 10: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for Sleep. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.68
Statistical Analysis 11: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for Enjoyment of Life. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.77
Statistical Analysis 12: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for BPI-I for Mean Interference Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.84

6. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity (CGI-S) at 8 Weeks
Description: The CGI-S scale evaluates the severity of illness at the time of assessment. The scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The CGI-S must be administered by a study physician in the presence of the participant or after having been in the presence of the participant. The Least Squares Mean estimates were adjusted for baseline, treatment, investigator (pooled), visit, treatment*visit, and baseline*visit.
Time Frame: Baseline, 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline CGI-S value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 244 | 247
units on a scale | -0.80 (0.07) | -1.16 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.35

7. Secondary Outcome: Change From Baseline in the Patient Global Assessment of Illness (PGAI) at 8 Weeks
Description: The PGAI is a participant-rated measure of the severity of osteoarthritis (OA) of the knee the participant has experienced in the past week as indicated on an 11-point numeric rating scale, with scores ranging from 0 to 10, where greater numbers reflect greater severity. The Least Squares Mean estimates were adjusted for baseline value, treatment, investigator (pooled), visit, treatment*visit, and baseline*visit.
Time Frame: Baseline, 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline PGAI value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 219 | 214
units on a scale | -1.77 (0.17) | -2.95 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -1.17

8. Secondary Outcome: Change From Baseline in the Profile of Mood States-Brief Form (BPOMS) Total and Subscale Scores at 8 Weeks
Description: 30-item BPOMS measures positive and negative aspects of mood states (item score: 0=not at all to 4=extremely). 5 negative factors: tension-anxiety, depression-dejection, anger-hostility, fatigue-inertia, confusion-bewilderment; 1 positive factor: vigor-activity. Factor scores range: 0 to 20; high scores=negative mood (positive mood for vigor). Total score=sum of 5 negative factor scores minus vigor score; range: -20=least disturbed to 100=most disturbed. Least Squares Mean estimates adjusted for baseline value, treatment, investigator (pooled), visit, treatment*visit, and baseline value*visit.
Time Frame: Baseline, 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline BPOMS value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 220 | 216
units on a scale
  BPOMS Total Score | -4.15 (0.89) | -4.98 (0.88)
  BPOMS Tension-Anxiety Score | -0.90 (0.21) | -1.17 (0.20)
  BPOMS Depression-Dejection Score | -0.51 (0.21) | -0.85 (0.20)
  BPOMS Anger-Hostility Score | -0.63 (0.21) | -1.15 (0.21)
  BPOMS Vigor-Activity Score | -0.34 (0.33) | 0.04 (0.32)
  BPOMS Fatigue-Inertia Score | -1.40 (0.30) | -1.47 (0.29)
  BPOMS Confusion-Bewilderment Score | -0.29 (0.17) | -0.32 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.449, Mixed Models Analysis — This is the p-value for the BPOMS Total Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.83
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.265, Mixed Models Analysis — This is the p-value for the BPOMS Tension-Anxiety Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.28
Statistical Analysis 3: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.180, Mixed Models Analysis — This is the p-value for the BPOMS Depression-Dejection Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.34
Statistical Analysis 4: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis — This is the p-value for the BPOMS Anger-Hostility Score. 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.52
Statistical Analysis 5: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.356, Mixed Models Analysis — This is the p-value for the BPOMS Vigor-Activity Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = 0.37
Statistical Analysis 6: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.862, Mixed Models Analysis — This is the p-value for the BPOMS Fatigue-Inertia Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.06
Statistical Analysis 7: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.883, Mixed Models Analysis — This is the p-value for the BPOMS Confusion-Bewilderment Score. A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -0.03

9. Secondary Outcome: Percentage of Participants Using Acetaminophen Weekly During the 10-Week Treatment Period
Description: The Least Squares (LS) Mean percentage estimates of participants using acetaminophen was determined during each week individually over the full 10-week treatment period based on participant's daily Yes/No assessments for the use of acetaminophen. The LS Mean estimates for the main effect of treatment (average weekly use) were adjusted for baseline value, treatment, investigator (pooled), week, and treatment*week.
Time Frame: Baseline through 10 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline weekly acetaminophen use value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 258 | 262
percentage of participants | 26 (2) | 22 (2)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.083, Mixed Models Analysis — A 0.05 level of significance was pre-specified for use in treatment group comparisons; In Mixed Models Analysis, degrees of freedom were estimated using the Kenward-Rogers approximation; Mean Difference (Final Values) = -4

10. Secondary Outcome: Percentage of Responders as Assessed by the Osteoarthritis Research Society International (OARSI) Response Criteria up to 8 Weeks
Description: OARSI response is composite Yes/No response assessed at 8 weeks based on decrease in 24-hour average pain ratings, range: 0 ("no pain") to 10 ("worst possible pain"), improvement in functioning (using WOMAC physical function scores, range: 0 [no difficulty] to 68 [extreme difficulty]), and improvement in participant's impression of illness (using PGAI scores, range: 0 to 10; 10=greatest severity). OARSI responder=large response in pain or function components (50% relative and 20% absolute improvement), or moderate response (20% relative and 10% absolute improvement) in 2 of 3 components.
Time Frame: Up to 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline OARSI response value, last-observation-carried forward (LOCF) based on values of each of the 3 components listed in the outcome measure description were included in the analysis.
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 259 | 263
percentage of responders | 48.3 | 69.6
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Fisher Exact — A 0.05 level of significance was pre-specified for use in treatment group comparisons

11. Secondary Outcome: Percentage of Participants Who Achieved a 30 Percent or 50 Percent Reduction in the Weekly Mean of the 24-Hour Average Pain Score up to 8 Weeks
Description: Response is a dichotomous outcome (Yes/No) indicating at least 30% (or 50%) reduction from baseline to endpoint for the weekly mean of the 24-hour average pain ratings. The weekly mean 24-hour average pain score was calculated from the participant's daily 24-hour average pain rating assessed on an 11-point numeric rating scale, with scores from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: Up to 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline weekly mean of the 24-hour average pain score value, last-observation-carried forward (LOCF) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 255 | 259
percentage of participants
  30% Response (LOCF) based on 24-Hour Average Pain | 33.7 | 53.7
  50% Response (LOCF) based on 24-Hour Average Pain | 16.1 | 35.5
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Fisher Exact — This is the p-value for the 30% Response (LOCF) based on 24-Hour Average Pain Ratings. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Fisher Exact — This is the p-value for the 50% Response (LOCF) based on 24-Hour Average Pain Ratings. A 0.05 level of significance was pre-specified for use in treatment group comparisons

12. Secondary Outcome: Percentage of Participants Who Achieved a 30 Percent or 50 Percent Reduction in the Brief Pain Inventory-Severity (BPI-S) Average Pain Score up to 8 Weeks
Description: Response is a dichotomous outcome (Yes/No) indicating at least 30% (or 50%) reduction from baseline to endpoint for BPI-S average pain rating. The BPI-S self-reported scale that measures the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Up to 8 weeks (blinded endpoint)
Population: Modified intent to treat (mITT) population: ITT participants with a baseline and at least 1 post-baseline BPI-S average pain value, last-observation-carried forward (LOCF) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 256 | 258
percentage of participants
  30% Response (LOCF) based on BPI-S Average Pain | 34.0 | 58.1
  50% Response (LOCF) based on BPI-S Average Pain | 21.1 | 45.7
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Fisher Exact — This is the p-value for the 30% Response (LOCF) based on BPI Average Pain Ratings
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p < 0.001, Fisher Exact — This is the p-value for the 50% Response (LOCF) based on BPI Average Pain Ratings

13. Other Pre Specified Outcome: Percentage of Participants With Abnormal High Hemoglobin A1c (HbA1c) up to 10 Weeks
Description: Abnormal high HbA1c is defined as a post-baseline HbA1c > 6.1% if baseline HbA1c ≤ 6.1% for lab samples obtained before November 17, 2010 and post-baseline HbA1c > 6.4% if baseline HbA1c ≤ 6.4% for lab samples obtained November 17, 2010 and beyond.
Time Frame: Up to 10 weeks
Population: Number of participants with a normal baseline and at least 1 post-baseline abnormal HbA1C value, last-observation-carried forward (LOCF) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 210 | 208
percentage of participants | 5.7 | 1.0
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.012, Fisher Exact — A 0.05 level of significance was pre-specified for use in treatment group comparisons

14. Other Pre Specified Outcome: Percentage of Participants With Abnormal Weight Gain and Weight Loss up to 10 Weeks
Description: Abnormal weight gain (potentially clinically significant [PCS] weight gain) is defined as weight gain at last visit ≥ 7% of the baseline weight.
  Abnormal weight loss (PCS weight loss) is defined as weight loss at last visit ≥ 7% of the baseline weight.
Time Frame: Up to 10 weeks
Population: Participants with a baseline and at least 1 post-baseline weight value, last-observation-carried forward (LOCF) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 256 | 258
percentage of participants
  PCS Weight Gain | 1.6 | 1.2
  PCS Weight Loss | 0.8 | 3.1
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.724, Fisher Exact — This is the p-value for PCS Weight Gain. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.106, Fisher Exact — This is the p-value for PCS Weight Loss. A 0.05 level of significance was pre-specified for use in treatment group comparisons

15. Secondary Outcome: Percentage of Participants Who Discontinued Due to an Adverse Event During the 10-Week Treatment Period
Time Frame: Baseline through 10 weeks
Population: All randomized participants were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 260 | 264
percentage of participants | 8.8 | 15.2
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.031, Fisher Exact — A 0.05 level of significance was pre-specified for use in treatment group comparisons

16. Other Pre Specified Outcome: Percentage of Participants With Abnormal Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) up to 10 Weeks
Description: Abnormal DPB (diastolic hypertension) is defined as sitting DBP ≥ 90 mm Hg that is also ≥ 10 mm Hg increase from baseline that is observed at last visit if highest baseline DBP < 90 mm Hg.
  Abnormal SBP (systolic hypertension) is defined as sitting SBP ≥ 140 mm Hg that is also ≥ 10 mm Hg increase from baseline that is observed at last visit if highest baseline SBP < 140 mm Hg.
Time Frame: Up to 10 weeks
Population: Participants with a normal baseline and at least 1 post-baseline DBP and SBP value, last-observation-carried forward (LOCF) were included in the analysis. Participants with a normal baseline value and a nonmissing endpoint value for the variable of interest were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 202 | 215
percentage of participants
  Diastolic Hypertension | 1.0 | 4.2
  Systolic Hypertension (N=170, 171) | 4.7 | 12.3
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.063, Fisher Exact — This is the p-value for Diastolic Hypertension. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.018, Fisher Exact — This is the p-value for Systolic Hypertension. A 0.05 level of significance was pre-specified for use in treatment group comparisons

17. Other Pre Specified Outcome: Percentage of Participants With Abnormal Pulse Rate up to 10 Weeks
Description: Abnormal pulse rate (tachycardia) is defined as a sitting heart rate (HR) ≥ 100 beats per minute (bpm) that is also ≥ 10 bpm compared to baseline, at last visit if highest baseline HR < 100 bpm.
Time Frame: Up to 10 weeks
Population: Participants with a normal baseline and at least 1 post-baseline pulse rate value, last-observation-carried forward (LOCF) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 257 | 264
percentage of participants | 0.0 | 1.1
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.249, Fisher Exact — A 0.05 level of significance was pre-specified for use in treatment group comparisons

18. Other Pre Specified Outcome: Percentage of Participants With a Change of Better, Worse, or No Change in Health Outcomes as Measured by Resource Utilization (REU) up to 10 Weeks
Description: REU captures information regarding the participant's work status and/or health care utilization. Investigators gather information from medical records, psychiatric history, and direct questioning of the participant and his or her family to complete the questionnaire. Responses to each item, comparing baseline to endpoint, are characterized as "Better," "Same," or "Worse." Better: an increase in time spent working/volunteering/holding a job, decrease in number of health care visits; Same: no change in time spent working/volunteering/holding a job, no change in number of health care visits; Worse: decrease in time spent working/volunteering/holding a job, increase in number of health care visits.
Time Frame: Up to 10 weeks
Population: Intent-to-treat (ITT) participants with a baseline and at least 1 post-baseline REU value, last-observation-carried forward (LOCF) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Duloxetine
Number analyzed (Participants) | 260 | 264
percentage of participants
  Outpatient Group Visits-Better | 0.4 | 0.0
  Outpatient Group Visits-Same | 99.6 | 100.0
  Outpatient Group Visits-Worse | 0.0 | 0.0
  Outpatient Individual Visits-Better | 2.4 | 0.8
  Outpatient Individual Visits-Same | 96.7 | 99.2
  Outpatient Individual Visits-Worse | 0.8 | 0.0
  ER Visits for Psychiatric Illness-Better | 0.0 | 0.0
  ER Visits for Psychiatric Illness-Same | 100.0 | 100.0
  ER Visits for Psychiatric Illness-Worse | 0.0 | 0.0
  ER Visits for Non-psychiatric Illness-Better | 5.7 | 3.7
  ER Visits for Non-psychiatric Illness-Same | 92.7 | 95.5
  ER Visits for Non-psychiatric Illness-Worse | 1.6 | 0.8
  Outpatient Visits to Other Physicians-Better | 20.4 | 26.0
  Outpatient Visits to Other Physicians-Same | 74.3 | 69.4
  Outpatient Visits to Other Physicians-Worse | 5.3 | 4.5
  Average Hours Worked for Pay per Week-Better | 15.2 | 18.9
  Average Hours Worked for Pay per Week-Same | 64.3 | 69.4
  Average Hours Worked for Pay per Week-Worse | 20.5 | 11.7
  How Long Participant Had This Job-Better | 25.2 | 20.2
  How Long Participant Had This Job-Same | 65.8 | 69.7
  How Long Participant Had This Job-Worse | 9.0 | 10.1
  Average Hours of Volunteer Work per Week-Better | 10.7 | 11.1
  Average Hours of Volunteer Work per Week-Same | 67.9 | 72.2
  Average Hours of Volunteer Work per Week-Worse | 21.4 | 16.7
  Psychiatric Visits-Better | 1.6 | 0.8
  Psychiatric Visits-Same | 98.4 | 99.2
  Psychiatric Visits-Worse | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.241, Likelihood Ratio Chi-squared — This is the p-value for outpatient group visits. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 2: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.087, Likelihood Ratio Chi-squared — This is the p-value for outpatient individual visits. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 3: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.414, Likelihood Ratio Chi-squared — This is the p-value for emergency room visits for non-psychiatric illness. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 4: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.332, Likelihood Ratio Chi-squared — This is the p-value for outpatient visits to other physicians. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 5: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.183, Likelihood Ratio Chi-squared — This is the p-value for the average number of hours worked for pay per week. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 6: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.666, Likelihood Ratio Chi-squared — This is the p-value for how long the participant has had this job. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 7: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.890, Likelihood Ratio Chi-squared — This is the p-value for the average number of hours of volunteer work per week. A 0.05 level of significance was pre-specified for use in treatment group comparisons
Statistical Analysis 8: Comparison: Placebo vs Duloxetine; Test type: Superiority or Other; p = 0.413, Likelihood Ratio Chi-squared — This is the p-value for psychiatric visits. A 0.05 level of significance was pre-specified for use in treatment group comparisons

ADVERSE EVENTS:
Arm/Group | Placebo | Duloxetine
Serious Adverse Events (participants affected / at risk) | 3/260 | 5/264
Other Adverse Events (participants affected / at risk) | 129/260 | 167/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=260) | Duloxetine (N=264)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=260) | Duloxetine (N=264)
Palpitations (Cardiac disorders) | 2 (2) | 4 (4)
Vision blurred (Eye disorders) | 1 (1) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 7 (7)
Constipation (Gastrointestinal disorders) | 8 (8) | 23 (24)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 18 (19)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 25 (25)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 12 (12) | 41 (43)
Vomiting (Gastrointestinal disorders) | 3 (3) | 11 (12)
Fatigue (General disorders) | 4 (4) | 18 (19)
Feeling jittery (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 3 (4) | 3 (3)
Therapeutic response unexpected (General disorders) | 4 (5) | 3 (4)
Thirst (General disorders) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (8) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2)
Liver function test abnormal (Investigations) | 0 (0) | 3 (3)
Weight increased (Investigations) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Dizziness (Nervous system disorders) | 7 (7) | 17 (17)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 10 (10) | 16 (21)
Somnolence (Nervous system disorders) | 7 (7) | 14 (14)
Tremor (Nervous system disorders) | 1 (1) | 3 (3)
Abnormal dreams (Psychiatric disorders) | 5 (5) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (5) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3) | 13 (15)
Libido decreased (Psychiatric disorders) | 1 (1) | 5 (5)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 6 (6)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (10)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days